CLINICAL TRIAL: NCT07388953
Title: Peripheral Autonomic Block (BAP) Plus Transversus Abdominis Plane Block (TAP) for Postoperative Analgesia After Minimally Invasive Left-Sided Colorectal Resection (BAPTAP): A Randomized, Controlled, Double-Blind Trial
Brief Title: Peripheral Autonomic Block (BAP) Plus Transversus Abdominis Plane Block (TAP) for Postoperative Analgesia After Minimally Invasive Left-Sided Colorectal Resection (BAPTAP)
Acronym: BAPTAP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Faculdade de Ciências Médicas de Minas Gerais (Other)
Collaborators: Santa Casa de Misericórdia de Belo Horizonte (Other)
Responsible Party: Principal Investigator, Alessandra Hubner de Souza, PhD, Faculdade de Ciências Médicas de Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 84933224.2.0000.5138
Record Dates: First submitted 2026-01-13; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Cancer; Colorectal Surgery; Anesthesia; Autonomic Nerve Block; Transversus Abdominis Plane (TAP) Block; Pain Management; Post Operative Analgesia
Keywords: colorectal surgery; Postoperative Pain; Peripheral Autonomic Block; Superior Hypogastric Plexus; Inferior Mesenteric Plexus; TAP Block; ERAS; Ropivacaine; Opioid-sparing Analgesia
MeSH Terms: conditions — Colorectal Neoplasms; Bites and Stings; Agnosia; Pain, Postoperative | interventions — Surgical Instruments

STUDY DESIGN:
Intervention Model Description: This is a single-center, individually randomized (1:1), two-arm, parallel-assignment, superiority trial. All participants receive standardized general anesthesia and perioperative ERAS care. Arm A (BAPTAP) receives a laparoscopic peripheral autonomic plexus block targeting the superior hypogastric and inferior mesenteric plexuses with ropivacaine 0.2% (8 mL per site) performed before dissection, plus a bilateral ultrasound-guided transversus abdominis plane (TAP) block with ropivacaine 0.33% (30 mL per side). Arm B (control) receives general anesthesia with trocar/wound infiltration only, without autonomic plexus or TAP blocks; postoperative analgesia follows the institutional ERAS protocol. Randomization occurs at the participant level with no crossover; the anesthesiologist performing the block is unblinded and is not involved is not involved in postoperative care or outcome assessments, while participants, and assessors remain masked.
Who Masked: Participant, Outcomes Assessor
Masking Description: andomization occurs at the participant level with no crossover; the anesthesiologist performing the block is unblinded and is not involved is not involved in postoperative care or outcome assessments, while participants, and assessors remain masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A - Experimental: BAPTAP (Peripheral Autonomic Block + TAP Block) (Experimental): General anesthesia and Peripheral autonomic plexus block (superior hypogastric and inferior mesenteric plexuses) with ropivacaine 0.2%, 8 mL per site; performed laparoscopically prior to dissection, associated with Bilateral ultrasound-guided TAP block using ropivacaine 0.33%, 30 mL per side.
  Interventions: Procedure: Minimally Invasive Left-Sided Colorectal Resection; Procedure: BAPTAP (Peripheral Autonomic Blockade + TAP Block)
- Arm B - Control: Trocar/wound infiltration (Standard of Care) (Active Comparator): General anesthesia and trocar/wound infiltration - ropivacaine 0.33% up to 60 mL total.
  Interventions: Procedure: Minimally Invasive Left-Sided Colorectal Resection; Procedure: Trocar/Incision Infiltration

INTERVENTIONS:
Procedure: Minimally Invasive Left-Sided Colorectal Resection — Elective laparoscopic anterior/rectosigmoid resection or sigmoid colectomy per institutional standards; not randomized.
Procedure: BAPTAP (Peripheral Autonomic Blockade + TAP Block) — General anesthesia combined with peripheral autonomic plexus blockade (superior hypogastric and inferior mesenteric plexuses) using 0.2% ropivacaine, 8 mL per site; performed laparoscopically prior to dissection, in association with bilateral ultrasound-guided TAP block with 0.33% ropivacaine, 30 mL per side.
  Arms: Arm A - Experimental: BAPTAP (Peripheral Autonomic Block + TAP Block)
Procedure: Trocar/Incision Infiltration — General anesthesia with trocar/incision infiltration using 0.33% ropivacaine, up to a total volume of 60 mL.
  Arms: Arm B - Control: Trocar/wound infiltration (Standard of Care)

SUMMARY:
Effective postoperative pain management is essential for enhanced recovery after laparoscopic colorectal surgery. This randomized, controlled, double-blind trial will compare conventional postoperative analgesia (intravenous medications plus surgical wound infiltration) with a locoregional strategy combining a peripheral autonomic block (inferior mesenteric and superior hypogastric plexuses) and a transversus abdominis plane (TAP) block. We hypothesize that the combined strategy (BAPTAP) reduces pain intensity and opioid consumption in the first 48 hours after Left-Sided Colorectal Resection.

DETAILED DESCRIPTION:
Postoperative pain after colorectal surgery involves both somatic and visceral components. Abdominal wall blocks target somatic nociception, whereas visceral pain often requires different approaches. Autonomic plexus blocks have shown promise in gynecologic and bariatric surgery. This study will randomize 140 adults undergoing elective laparoscopic Left-Sided Colorectal Resection to either: (1) BAPTAP (peripheral autonomic plexus block targeting the superior hypogastric and inferior mesenteric plexuses plus bilateral ultrasound-guided TAP block) in addition to standardized multimodal analgesia; or (2) Control (standardized multimodal analgesia and trocar/wound infiltration alone). Primary outcomes are pain intensity (Numerical Rating Scale) at predefined time points and cumulative opioid consumption (IV morphine equivalents) in the first 48 hours. Secondary outcomes include functional recovery milestones, adverse events, complications related to blocks or systemic analgesia, patient satisfaction, and quality of recovery via the PAIN OUT questionnaire. Randomization is computer-generated (1:1). Participants, postoperative care teams, and outcome assessors will be blinded; the anesthesiologist performing the block will not participate in postoperative assessments.

This is an interventional, randomized (1:1), parallel-assignment, double-masked clinical trial with an estimated enrollment of 140 participants, designed for supportive care (postoperative analgesia) in patients undergoing minimally invasive left-sided colorectal surgery for indications including colorectal neoplasms and diverticular disease, with outcomes focused on postoperative pain. Participants aged 18-80 years of any sex, ASA I-II, scheduled for elective laparoscopic Left-Sided Colorectal Resection at a single institution and able to understand and sign informed consent are eligible. Exclusions include known allergy to study medications (Ropivacaine), coagulation disorders, pregnancy, inability to provide consent, chronic pain on opioid therapy, and BMI > 35 kg/m². Two arms will be compared: the experimental arm receives a peripheral autonomic plexus block (targeting the superior hypogastric and inferior mesenteric plexuses) with ropivacaine 0.2% at 8 mL per site performed laparoscopically before dissection plus a bilateral ultrasound-guided TAP block with ropivacaine 0.33% at 30 mL per side, in addition to standard multimodal analgesia; the active comparator arm receives the same multimodal analgesia with trocar/wound infiltration using ropivacaine 0.33% up to 60 mL total, without autonomic plexus or TAP blocks. Masking is double (participant and outcomes assessor); the anesthesiologist who performs the block is unblinded and does not take part in postoperative care or assessments, while participants, and assessors remain blinded. The coprimary outcomes are pain intensity at rest on an NRS 0-10 at 2, 6, 12, 24, and 48 hours after surgery and cumulative opioid consumption over the first 48 hours expressed as intravenous morphine equivalents calculated as (fentanyl mg × 100) + (morphine IV mg) plus, if applicable, (tramadol mg ÷ 10); secondary outcomes include time to return of bowel function (first flatus and first bowel movement) through discharge, time to ambulation up to 48 hours, length of hospital stay during the index admission, adverse events and complications related to the TAP/autonomic blocks or systemic analgesia from the intraoperative period to 30 days postoperatively, patient-reported outcomes at 48 hours using PAIN OUT (Portuguese-validated IPO) covering pain frequency, interference with activities and mood, satisfaction, and participation, and overall patient satisfaction with pain management at 48 hours; an exploratory outcome consists of a 5-10 minute qualitative interview at 48 hours addressing expectations, trust, coping, and emotional impact.

ELIGIBILITY:
Inclusion Criteria:

* Elective laparoscopic left-sided colorectal resection
* ASA physical status I-II
* Ability to understand the study and sign informed consent

Exclusion Criteria:

* Known allergy to study medications (e.g., local anesthetics)
* Coagulation disorders
* Pregnancy
* Inability to understand or provide consent
* Chronic pain on opioid therapy
* BMI > 35 kg/m²

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2026-02-14 (Estimated); Primary Completion 2026-12-05 (Estimated); Study Completion 2027-07-05 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Day 0, day 1 and day 2 - From the surgical procedure up to 48 hours postoperatively
  Pain intensity at rest (NRS 0-10); Time Frame: 2 hours, 6 hours, 12 hours, 24 hours and 48 hours postoperatively; Higher scores indicate worse pain.
Cumulative opioid consumption | Day 0, day 1 and day 2 - From the surgical procedure up to 48 hours postoperatively
  Cumulative opioid consumption (IV morphine equivalents, mg) in the first 48 hours; Time Frame: baseline to 48 hours; Calculated as: (Fentanyl mg × 100) + (Morphine IV mg) [+ (Tramadol mg ÷ 10) if applicable].
Pain frequency - Patient-reported outcomes via PAIN OUT (Portuguese-validated IPO) | Day 2 - 48 hours postoperatively
  Pain frequency is assessed by evaluating both intensity and temporal occurrence of postoperative pain. Patients are asked to report:
  The worst pain intensity experienced since surgery, measured on an 11-point Numeric Rating Scale (NRS), ranging from 0 (no pain) to 10 (worst pain imaginable).
  The least pain intensity experienced during the same period, using the same scale.
  The frequency of severe pain, expressed as the estimated percentage of time the patient experienced severe pain since surgery, ranging from 0% (never) to 100% (always).
  This domain captures not only peak pain intensity but also pain variability and persistence over time.
Patient-reported outcomes via PAIN OUT (Portuguese-validated IPO) - interference with activities and mood | Day 2 - 48 hours postoperatively
  This domain evaluates the functional and emotional impact of postoperative pain.
  Interference with physical activities is assessed using an 11-point NRS (0 = did not interfere; 10 = completely interfered) in relation to:
  * Activities in bed (e.g., turning, sitting up, changing position)
  * Deep breathing or coughing
  * Sleep quality
  * Activities out of bed (e.g., walking, standing, sitting in a chair), when applicable
  Interference with mood and emotional well-being is evaluated by assessing the extent to which pain caused the patient to feel:
  * Anxious
  * Helpless
  Each emotional parameter is rated on an 11-point NRS from 0 (not at all) to 10 (extremely), reflecting the psychological burden associated with postoperative pain.
Participation - Patient-reported outcomes via PAIN OUT (Portuguese-validated IPO) | Day 2 - 48 hours postoperatively
  Participation assesses the patient's involvement in pain management decisions and information exchange. It includes:
  The degree to which the patient felt allowed to participate in decisions regarding pain treatment, rated on an 11-point NRS from 0 (not at all) to 10 (very much so).
  Whether the patient received information about available pain treatment options (yes/no).
  Whether the patient would have preferred more pain treatment than was provided (yes/no).
  This domain emphasizes shared decision-making, patient autonomy, and communication quality within postoperative pain management.

SECONDARY OUTCOMES:
Patient satisfaction with pain management | Day 2 - 48 hours postoperatively
  Patient satisfaction with pain management is assessed through two complementary measures: Overall satisfaction with pain treatment outcomes, rated on an 11-point NRS ranging from 0 (extremely dissatisfied) to 10 (extremely satisfied). Perceived adequacy of pain relief, expressed as a percentage from 0% (no relief) to 100% (complete relief), considering all pain treatments combined (pharmacological and non-pharmacological). This domain reflects the patient's global evaluation of analgesic effectiveness and quality of care.
Time to return of bowel function | From D0 up to 1 month
  Time to return of bowel function was defined as the interval, in hours, from the end of the surgical procedure to the recovery of gastrointestinal motility.
  Outcome Components
  The return of bowel function was assessed based on the following clinical parameters:
  * Time to first passage of flatus
  * Time to first bowel movement (defecation)
Length of hospital stay. | Day 30
  Length of hospital stay; Time Frame: index admission
Time to ambulation. | Day 0, day 1 and day 2 - from the surgical procedure up to 48 hours postoperatively
  Time to ambulation; Time Frame: up to 48 hours.
Adverse events and complications related to TAP/BAP/systemic analgesia. | Day 30

OTHER OUTCOMES:
Qualitative interview (5-10 min) on expectations, trust, coping, and emotional impact. | Day 2 - 48 hours postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Santa Casa de Misericórdia de Belo Horizonte, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: Yes
We plan to share de-identified individual participant data (IPD) underlying the primary and secondary outcomes of this trial, including demographics, intraoperative variables necessary to interpret outcomes, postoperative pain scores at prespecified time points, cumulative opioid use (IV morphine equivalents), adverse events, length of stay, and discharge status. Direct identifiers and free-text notes will be removed; a re-identification key will be retained only at the site and will not be shared. Accompanying documents (final protocol, statistical analysis plan, data dictionary/codebook, blank CRFs, informed consent template, and analytic code for the primary analyses) will be provided. Access will be granted to qualified researchers with a methodologically sound proposal and IRB/ethics approval (or exemption) who sign a data-use agreement compliant with Brazil's LGPD (Law No. 13,709/2018) and institutional policies. Requests should be sent to the corresponding author.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available beginning 6 months after publication of the primary results for 36 months (extensions considered upon reasonable request).
Access Criteria: Access will be granted to qualified researchers with a methodologically sound proposal and IRB/ethics approval (or exemption) who sign a data-use agreement compliant with Brazil's LGPD (Law No. 13,709/2018) and institutional policies.

REFERENCES:
- [Background] Daes J, Morrell DJ, Hanssen A, Caballero M, Luque E, Pantoja R, Luquetta J, Pauli EM. Paragastric Autonomic Neural Blockade to Prevent Early Visceral Pain and Associated Symptoms After Laparoscopic Sleeve Gastrectomy: a Randomized Clinical Trial. Obes Surg. 2022 Nov;32(11):3551-3560. doi: 10.1007/s11695-022-06257-9. Epub 2022 Sep 2. PMID 36050617
- [Background] Diaz-Cambronero O, Mazzinari G, Cata JP. Perioperative opioids and colorectal cancer recurrence: a systematic review of the literature. Pain Manag. 2018 Sep 1;8(5):353-361. doi: 10.2217/pmt-2018-0029. Epub 2018 Sep 13. PMID 30212256
- [Background] Zeng J, Hong A, Gu Z, Jian J, Liang X. Efficacy of transversus abdominis plane block on postoperative nausea and vomiting: a meta-analysis of randomized controlled trial. BMC Anesthesiol. 2024 Mar 1;24(1):87. doi: 10.1186/s12871-024-02469-x. PMID 38429757
- [Background] Urits I, Schwartz R, Herman J, Berger AA, Lee D, Lee C, Zamarripa AM, Slovek A, Habib K, Manchikanti L, Kaye AD, Viswanath O. A Comprehensive Update of the Superior Hypogastric Block for the Management of Chronic Pelvic Pain. Curr Pain Headache Rep. 2021 Feb 25;25(3):13. doi: 10.1007/s11916-020-00933-0. PMID 33630172
- [Background] Lopez-Ruiz C, Orjuela JC, Rojas-Gualdron DF, Jimenez-Arango M, Rios JFL, Vasquez-Trespalacios EM, Vargas C. Efficacy of Transversus Abdominis Plane Block in the Reduction of Pain and Opioid Requirement in Laparoscopic and Robot-assisted Hysterectomy: A Systematic Review and Meta-analysis. Rev Bras Ginecol Obstet. 2022 Jan;44(1):55-66. doi: 10.1055/s-0041-1740595. Epub 2022 Jan 29. PMID 35092960
- [Background] De Silva P, Daniels S, Bukhari ME, Choi S, Liew A, Rosen DMB, Conrad D, Cario GM, Chou D. Superior Hypogastric Plexus Nerve Block in Minimally Invasive Gynecology: A Randomized Controlled Trial. J Minim Invasive Gynecol. 2022 Jan;29(1):94-102. doi: 10.1016/j.jmig.2021.06.017. Epub 2021 Jun 29. PMID 34197956
- [Background] De Pinto M, Cahana A. Medical management of acute pain in patients with chronic pain. Expert Rev Neurother. 2012 Nov;12(11):1325-38. doi: 10.1586/ern.12.123. PMID 23234394
- [Background] Baeriswyl M, Zeiter F, Piubellini D, Kirkham KR, Albrecht E. The analgesic efficacy of transverse abdominis plane block versus epidural analgesia: A systematic review with meta-analysis. Medicine (Baltimore). 2018 Jun;97(26):e11261. doi: 10.1097/MD.0000000000011261. PMID 29952997
- [Background] Aytuluk HG, Kale A, Basol G. Laparoscopic Superior Hypogastric Blocks for Postoperative Pain Management in Hysterectomies: A New Technique for Superior Hypogastric Blocks. J Minim Invasive Gynecol. 2019 May-Jun;26(4):740-747. doi: 10.1016/j.jmig.2018.08.008. Epub 2018 Aug 28. PMID 30165185